CLINICAL TRIAL: NCT03570710
Title: Reducing Blood Loss During Cesarean Hysterectomy for Placenta Accreta Spectrum With Intravenous Versus Topical Tranexamic Acid: A Double-blind Randomized Controlled Trial
Brief Title: Reducing Blood Loss During Cesarean Hysterectomy for Placenta Accreta Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/183/10/17
Record Dates: First submitted 2018-05-14; First posted 2018-06-27 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; placenta accreta spectrum; tranexamic acid
MeSH Terms: conditions — Placenta Accreta | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Eligible participants were allocated to one of three groups. Group (I): patients received 110 ml normal saline IV just before skin incision Group (II): patients received 1 gm TA (2 ampoules of Capron 500 mg /5 ml; Amoun, Cairo, Egypt) intravenous just before skin incision. Group (III): patients received 2 gm topical TA (4 ampoules of Capron 500 mg/5 ml) applied on the placental bed after placental delivery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- normal saline arm group (Placebo Comparator): 110 ml normal saline IV just before skin incision plus topical application of 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy
  Interventions: Drug: Normal saline
- intravenous tranexamic acid group (Active Comparator): 1 gm tranexamic acid (2 ampoules of Capron 500 mg /5 ml; Amoun, Cairo, Egypt) intravenous just before skin incision plus110 ml normal saline IV just before skin incision plus topical application of 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy
  Interventions: Drug: intravenous tranexamic acid
- Topical tranexamic acid group (Active Comparator): 2 gm topical tranexamic acid ( 4 ampoules of Capron 500 mg/5 ml applied typically) in 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy plus110 ml normal saline IV just before skin incision plus topical application of 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy plus In topical tranexamic acid group gauze soaked with 2g tranexamic acid (20 ml) diluted in 200 ml of sodium chloride 0.9% or placebo (120ml of sodium chloride 0.9%.) applied on the pelvic bed after Cesarean hysterectomy. To ensure a sufficiently high concentration, the tranexamic acid was diluted only to a volume sufficient to moisten a large wound surface. 20 ml moisten at least 1500 cm2.
  Interventions: Drug: Topical tranexamic acid

INTERVENTIONS:
Drug: intravenous tranexamic acid — 1 gm tranexamic acid (2 ampoules of Capron 500 mg /5 ml; Amoun, Cairo, Egypt) intravenous just before skin incision plus110 ml normal saline IV just before skin incision plus topical application of 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy
  Other Names: Active Comparator
  Arms: intravenous tranexamic acid group
Drug: Topical tranexamic acid — 2 gm topical tranexamic acid ( 4 ampoules of Capron 500 mg/5 ml applied typically) in 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy plus110 ml normal saline IV just before skin incision plus topical application of 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy plus In topical tranexamic acid group gauze soaked with 2g tranexamic acid (20 ml) diluted in 200 ml of sodium chloride 0.9% or placebo (120ml of sodium chloride 0.9%.) applied on the pelvic bed after Cesarean hysterectomy. To ensure a sufficiently high concentration, the tranexamic acid was diluted only to a volume sufficient to moisten a large wound surface. 20 ml moisten at least 1500 cm2.
  Other Names: Active Comparator
  Arms: Topical tranexamic acid group
Drug: Normal saline — 110 ml normal saline IV just before skin incision plus topical application of 200 ml normal saline applied on the pelvic bed after Cesarean hysterectomy
  Other Names: Placebo Comparator
  Arms: normal saline arm group

SUMMARY:
PAS is an obstetrics condition that is closely linked with massive obstetrical hemorrhage with a varied incidence about once in every 533 live births. It is considered one of the causes of massive transfusion (>4 units of packed red blood cells) and cesarean hysterectomy.

It is estimated that peripartum hysterectomies are performed in approximately0.08% of all deliveries. A large study from the United Kingdom noted that 38% were a result of PAS. More recently, population-based analyses show that PAS is the indication for the majority of peripartum hysterectomies.

Bleeding at the time of peripartum hysterectomy for PAS is often substantial. Nearly 90% of patients need blood products, while 38% of patients need a massive blood transfusion.

There is a 30% risk of an ICU admission, thromboembolic disease, readmission, reoperation, poor wound healing, and a reported rate of surgical re-exploration ranging from 4% to 33%. The risk of maternal death reported being as high as 7% (although less in most recent series) Therefore, adequate homeostatic techniques are essential. Currently, surgical hemostasis can be secured by a variety of methods, including mechanical sutures (or clamping), electric coagulation, ultrasonically activated scalpel or drugs.

TA is a lysine analog which acts as an antifibrinolytic via competitive inhibition of the binding of plasmin and plasminogen to fibrin. The rationale for its use in the reduction of blood loss depending on the implication of the coagulation and fibrinolysis processes . However, concerns about possible thromboembolic events with the parental administration of TA has stimulated increasing interest in its topical Use

DETAILED DESCRIPTION:
Eligible participants were allocated to one of three groups. Group (I): patients received 110 ml normal saline IV just before skin incision Group (II): patients received 1 gm TA (2 ampoules of Capron 500 mg /5 ml; Amoun, Cairo, Egypt) intravenous just before skin incision. Group (III): patients received 2 gm topical TA (4 ampoules of Capron 500 mg/5 ml) applied on the placental bed after placental delivery. Patients were randomized to three groups, each compromised of 43 patients according to a three-blocked randomization list which was coded (1 or 2 or 3) at 1:1:1 ratio. The three parallel groups were prepared using a Computer-generated randomization system. The allocated groups will be concealed in serially numbered sealed opaque envelopes that will only be opened after recruitment. The patient allocation will be performed prior to the induction of anesthesia by an independent person, who will not otherwise be involved in this study. The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used. In all eligible participants, CH was performed under general anesthesia by the same operative and anesthesia team. A dose of 1 g of first-generation cephalosporin (Cefazolin®; Bristol Mayers Squibb, Cairo, Egypt) was administered intravenously immediately prior to skin incision. The abdomen was exposed through Pfannensteil incision. After skin incision, the subcutaneous fat and abdominal fascia were opened crosswise, and the rectus muscle was opened on the midline, the parietal peritoneum was opened longitudinally, the visceral peritoneum was opened transversely and dissected downwards with the bladder and kept against symphysis pubis by a Doyen retractor, followed by transverse incision of the uterus at the upper border of the placenta to avoid transplacental incision which provoke severe bleeding.

Eligible participants were allocated to one of three groups after induction of general anesthesia and immediately prior to the operation and just before skin incision. they received 1-gram tranexamic acid (10 ml) in 100 ml saline infusion or placebo (110 normal saline) by slow intravenous injection at an approximate rate of 1 mL per min. Throughout the operation irrigation was done by 60 ml of (2g tranexamic acid (10 ml) diluted in 100 ml of sodium chloride 0.9%) or placebo ( 60 ml of sodium chloride 0.9%.).At the end of operation another dose of 60 ml of (1g tranexamic acid (10 ml) diluted in 50 ml of sodium chloride 0.9%) or placebo ( 60 ml of sodium chloride 0.9%.) was left intraabdominal then 1 intraperitoneal suction drain was routinely used in all patients the drains were closed for 3 hour postoperative , after that time the drains were opened and removed on the second postoperative day unless otherwise indicated.. To ensure a sufficiently high concentration of topical tranexamic acid, it was diluted only to a volume sufficient to moisten a large wound surface. 20 ml moistens at least 1500 cm2.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women with a single fetus scheduled for elective cesarean hysterectomy for placenta accreta spectrum

Exclusion Criteria:

* Patients with a cardiac, hepatic, renal or thromboembolic disease.
* patients with pelvic endometriosis and adnexal mass.
* patients had an allergy to tranexamic acid.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
intraoperative blood loss | during the operation
  intraoperative blood loss

SECONDARY OUTCOMES:
postoperative blood loss | 6 hours post operative
  postoperative blood loss
blood transfusion | intraoperative and 12 hour post operative
  intraoperative and 12 hour post operative

CONTACTS AND LOCATIONS:
Locations (1):
- AswanUH, Aswān, Egypt